CLINICAL TRIAL: NCT06345352
Title: Evaluation of the Quality of Care in the Emergency Department by Studying the Appropriateness of the Admissions of Patients Accessing the PS: Construction and Validation of an Algorithm Based on Computerised Databases
Brief Title: Evaluation of the Quality of Care in the Emergency Department by Studying the Appropriateness of Admissions of Patients Accessing the Emergency Department (Fondazione IRCCS Ca' Granda Ospedale Maggione Policlinico)
Status: Active, not recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: IRFMN_7520_PoliMI
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Quality of Care; Evaluation; Emergency Department; Appropriateness
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elegible population: All adult patients presenting to the emergency department with non-specific cardiopulmonary or abdominal manifestations, represented by one or more of the following symptoms: chest pain, abdominal pain, dyspnoea, transient loss of consciousness.

SUMMARY:
The aim of this study is to develop, study and validate a rigorous and sustainable method for assessing the clinical appropriateness of the decision taken in the Emergency Department to admit or not to admit patients.

DETAILED DESCRIPTION:
The information normally recorded in the Emergency Department medical record will be used, as well as the available clinical and administrative databases. For reasons of feasibility, the investigators will also restrict the analysis to patients coming to the Emergency Department with non-specific manifestations in the pulmonary, cardiovascular and abdominal districts, represented by one or more of the following symptoms: dyspnoea, chest pain, transient loss of consciousness, abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Presentation in the Emergency Department with non-specific cardiopulmonary or abdominal manifestations, represented by one or more of the following symptoms: chest pain, abdominal pain, dyspnoea, transient loss of consciousness.

Exclusion Criteria:

* Voluntary removal of the patient;
* Sending home with instructions to return for further services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients entering Emergency Department represented by one or more of the following symptoms: chest pain, abdominal pain, dyspnoea, transient loss of consciousness.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Algorithm creation | September 2020 - January 2024
  To develop, for the types of patients taken into consideration, a classification algorithm of the appropriateness of admissions based on the files available at the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico (for simplicity: Policlinico hospital)
Algorithm validation | February 2024 - December 2024
  To validate the classification algorithm on a sample of hospital medical records.
Algorithm application | January 2025 - December 2027
  To apply the validated algorithm on patients referred to the PS of the Policlinico hospital over 36 months, to estimate the proportion of appropriate admissions.
Appropriateness estimation | January 2025 - December 2027
  Provide, for the types of patients considered, an estimate of appropriate discharges for patients discharged and subsequently admitted to the Polyclinic, by drawing on the data available at the polyclinic itself. For all other patients, data on living status and admissions to other facilities in the metropolitan area (PS administrative flow and hospital discharge cards - SDOs), will be analysed using data provided by the ATS Milano Città Metropolitana.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided